CLINICAL TRIAL: NCT05952609
Title: A 2-year Clinical Performance of Two Different Ion-releasing Bulk-fill Restorative Materials Placed in Posterior Cavities
Brief Title: A 2-year Clinical Performance of Two Different Ion-releasing Bulk-fill Restorative Materials Posterior Cavities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M02060421
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2021-04

CONDITIONS: Secondary Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Patients receiving Surefil One
  Interventions: Other: Surefil One
- Group 2 (Experimental): Patients receiving Cention N
  Interventions: Other: Cention N
- Group 3 (Active Comparator): Patients receiving bulkfil resin composite
  Interventions: Other: Bulkfil resin composite

INTERVENTIONS:
Other: Surefil One — Ion-releasing restoration
  Arms: Group 1
Other: Cention N — Ion-releasing restoration
  Arms: Group 2
Other: Bulkfil resin composite — resin composite (No ion-release)
  Arms: Group 3

SUMMARY:
The aim of this study is to evaluate and compare the clinical performance of 2 ion-releasing bulk-fill restorative materials in comparison with a bulk-fill resin composite restoration in posterior cavities.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for patient's inclusion in the study will be the presence of at least 3 occlusal or proximal carious lesion in posterior teeth, favourable and stable occlusion between the remaining teeth, the patients must be older than 18 years old with permanent dentition, moderate oral hygiene, asymptomatic vital teeth with no sensitivity to percussion, and the presence of contact with adjacent teeth

Exclusion Criteria:

* Exclusion criteria will be, sever bruxism, patients with known unavailability to attend recall visits, patients with known allergy to any component of the study materials, pulp exposure during caries excavation, patients with unstable medical conditions and pregnant or lactating individuals.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Evaluating surface and marginal staining | 2 years
  FDI criteria will be used
Evaluating fracture and retention of the materials | 2-years
  FDI criteria will be used
Evaluating marginal adaptation and discoloration of the materials | 2-years
  FDI criteria will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlyia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided